CLINICAL TRIAL: NCT02553447
Title: A Pilot Study of Vitamin D Replacement in Patients With Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia With Low Vitamin D Levels
Brief Title: Cholecalciferol in Newly Diagnosed Non-Hodgkin Lymphoma or Chronic Lymphocytic Leukemia With Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0556-15-FB; NCI-2015-01502 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma; Untreated Chronic Lymphocytic Leukemia; Vitamin D Deficiency
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (high-dose cholecalciferol) (Experimental): Patients receive high-dose cholecalciferol PO daily for 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis
- Arm II (low-dose cholecalciferol) (Experimental): Patients receive low-dose cholecalciferol PO daily for 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis
- Arm III (control) (No Intervention): Patients receive no intervention.

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
  Arms: Arm I (high-dose cholecalciferol); Arm II (low-dose cholecalciferol)
Other: Laboratory Biomarker Analysis — Optional correlative studies
  Arms: Arm I (high-dose cholecalciferol); Arm II (low-dose cholecalciferol)

SUMMARY:
This randomized pilot early phase I trial studies how well cholecalciferol works in treating patients with newly diagnosed non-Hodgkin lymphoma or chronic lymphocytic leukemia with low levels of vitamin D (vitamin D deficiency). Cholecalciferol may increase levels of vitamin D and improve survival in patients with non-Hodgkin lymphoma or chronic lymphocytic leukemia receiving standard of care chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 3 year progression-free survival (PFS), defined as time from the time of study entry of watch and wait or newly diagnosed non-Hodgkin lymphoma (NHL) or chronic lymphocytic leukemia (CLL) until relapse, progression, or death from any cause.

SECONDARY OBJECTIVES:

I. To evaluate changes in the levels of serum vitamin D levels during therapy with daily oral vitamin D supplementation (cholecalciferol).

II. To evaluate the overall survival (OS), defined as time from the time of study entry of watch and wait patients or newly diagnosed NHL or CLL until death from any cause.

OUTLINE: Patients with low levels of vitamin D are randomized to 1 of 2 arms and patients with normal levels are assigned to Arm III.

ARM I: Patients receive high-dose cholecalciferol orally (PO) daily for 3 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive low-dose cholecalciferol PO daily for 3 years in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed newly diagnosed or previously untreated (patients may be under no treatment ?wait and watch? or have received two cycles of chemotherapy or localized radiation therapy before going on this study) non-Hodgkin?s lymphoma or CLL
* Patients must have serum 25-hydroxyvitamin D (25[OH]D) drawn at time of enrollment; (NOTE: subjects currently taking vitamin D supplements are eligible for screening)
* Simultaneous participation in other therapeutic clinical trials will be allowed
* Patients must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* History of uncontrollable allergic reactions to vitamin D
* History of Paget?s disease
* Hypercalcemia
* Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the investigator?s opinion, may interfere with protocol adherence or a subject?s ability to give informed consent
* Inability to cooperate with the requirements of the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Time from the time of study entry of watch and wait or diagnosed non-Hodgkin lymphoma or chronic lymphocytic leukemia until relapse, progression, or death from any cause, assessed at 3 years
  The 3-year progression-free survival will be presented using Kaplan-Meier curves and will be presented for the normal serum vitamin D control group and the low and high dose randomized groups. Each randomized group (low and high dose) will be compared to a historical fixed expected 3-year progression-free survival of 45% using a one-sample logrank test following the method of Woolson (1981).

SECONDARY OUTCOMES:
Incidence of adverse events and serious events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days
  Will be described for the low dose and high dose groups and compared between groups using a Chi-square. The frequency of occurrence of overall toxicity, categorized by toxicity grades, will be described for the low dose and high dose groups and compared between groups using a Chi-square.
Overall survival | Time from the time of study entry of watch and wait or newly diagnosed non-Hodgkin lymphoma or chronic lymphocytic leukemia administered on trial until death from any cause, assessed at 3 years
  The 3-year overall survival will be presented using Kaplan-Meier curves and will be presented for the normal serum vitamin D control group and the low and high dose randomized groups. Each randomized group (low and high dose) will be compared to a historical fixed expected 3-year overall survival of 80% using a one-sample logrank test following the method of Woolson (1981).

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, MBA, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States